CLINICAL TRIAL: NCT05731752
Title: Phase I Clinical Trial of Tolerability and Pharmacokinetics of HX009 in Patients With Advanced Solid Tumors
Brief Title: Study on the Tolerability and Pharmacokinetics of HX009 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Hanx Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX009-I-01(CN)
Record Dates: First submitted 2023-01-29; First posted 2023-02-16 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX009 (Experimental): Study treatment: HX009 administered every 2 weeks (14 [±3] days) via intravenous infusion.
  Interventions: Drug: HX009

INTERVENTIONS:
Drug: HX009 — The subjects will receive HX009 treatment via IV infusion once every 2 weeks at different dose escalation cohorts
  Other Names: Recombinant humanized anti-CD47/PD-1 bifunctional antibody

SUMMARY:
This is an open, multiple-dose administration dose exploratory clinical phase I study to evaluate the safety, tolerability, and PK profile of HX009 Injection in patients with advanced solid tumors and to provide a preliminary measure of its antitumor efficacy. It includes Phase Ia and Phase Ib.

phase Ia is a dose exploratory study to evaluate safety, tolerability, and to determine the MTD and/or RP2D.The sponsor and investigator will adjust the magnitude of the dose escalation and the dosing cycle based on the safety and tolerability of HX009 Injection and the PK data that have been obtained, as well as decide whether to add an unplanned dose or dosing cycle to the trial, and recommend the RP2D.The Ia phase dose escalation design model is shown below. The planned dosing cycle for this study is once every 2 weeks (14 days) (Q2W) with IV HX009.

Based on the result of phase 1a,10 mg/kg Q2W was the recommended dose for phase 1b. The aimed population for 1b is patients diagnosed with advanced melanoma, and divided into two cohorts:: cohort A ,untreated patients with unresectable or metastatic advanced melanoma;and Cohort B, patients with unresectable or metastatic malignant melanoma that had been treated with immune checkpoint inhibitor therapy. The enrollment of Cohort B will start first.,and whether the cohort A will be initiated depends on the results of the cohort B .The up to 80 patients will be enrolled in Phase Ib.

DETAILED DESCRIPTION:
The study is divided into a screening, treatment, and follow-up period. The Treatment Period may continue to be administered until the investigator determines that the subject no longer benefits, or the subject develops intolerable toxicity, or the subject withdraws informed consent, or the disease progresses or is treated with an antineoplastic agent other than those specified in the protocol, or the subject dies, or is lost to follow-up, or a Phase Ib subject has been administered for 2 years (whichever occurs earliest).

Subjects who withdraw from the study/terminate treatment for any reason are required to return for 1 follow-up visit after the last dose, to collect as many RO blood samples as possible after discontinuation (only partial subjects in Phase Ib), and to collect clinical data on safety as well as survival. During the subsequent follow-up period (for Phase Ib only), subjects or family members will receive a telephone visit to inquire about survival and antitumor therapy.

ELIGIBILITY:
Inclusion Criteria:

In Phase Ia.

Subjects must meet all of the following enrollment criteria to be enrolled in this study:

1. Voluntarily sign an informed consent form, understand the study and be willing to follow and be capable of completing all trial procedures;
2. Male or female, age 18-70 years (including borderline values);
3. ECOG score: 0 to 1;
4. Advanced malignant solid tumors diagnosed by cytology or histopathology and after failure of standard treatment (disease progression or intolerable) or in the absence of effective therapies;
5. Subjects must have at least one extracranial lesion for efficacy assessment according to the Solid Tumor Evaluation Criteria (RECIST 1.1), including both measurable and non-measurable lesions. The number of subject cases with all non-measurable lesions must not exceed 1/3 of the total enrollment;
6. Expected survival ≥ 12 weeks;
7. If prior antitumor therapy has been received, the following are required:

   * ≥ 3 weeks between systemic radiation therapy and the first dose, and ≥ 2 weeks between localized radiation therapy or radiation therapy for bone metastases;
   * Prior chemotherapy, immunotherapy (PD-1 antibody, PD-L1 antibody, or CTLA-4 antibody, etc.), biologic therapy (tumor vaccine, cytokine, or growth factor for cancer control), and targeted therapy ≥ 4 weeks from the first administration interval (small molecule targeted agent therapy ≥ 2 weeks from the first administration interval);
   * Prior immunotherapy with PD-1 antibody, PD-L1 antibody, or CTLA-4 antibody without permanent discontinuation due to prior immunotherapy;
   * Prior treatment with a significant anti-tumor herbal or proprietary Chinese medicine ≥ 2 weeks from the first dose;
8. In the case of patients with asymptomatic Central Nervous System (CNS) metastases or treated asymptomatic brain metastases, be free of disease progression by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI), be stable for at least 4 weeks, and not require steroid medication;
9. Have appropriate organ and hematopoietic function and no severe cardiac, pulmonary, hepatic, or renal dysfunction or immunodeficiency based on the following laboratory tests

in phase Ib

Subjects must meet all of the following enrollment criteria to be enrolled in this trial:

1. Voluntarily sign an informed consent form, understand the study and be willing to follow and be capable of completing all trial procedures;
2. Male or female, age 18-75 years (including borderline values);
3. ECOG score: 0 to 1;
4. Unresectable/metastatic advanced melanoma diagnosed by cytology or histopathology;
5. Cohort A: No prior systemic therapy for advanced melanoma (prior neoadjuvant and adjuvant therapy with last dose completed before 6 months can be enrolled). Cohort A: No prior systemic therapy for advanced melanoma (previous neoadjuvant and adjuvant therapy, completed before 6 months of last dose) Cohort B: Disease progression after treatment with immune checkpoint inhibitors ;
6. Subjects must have at least one measurable lesion according to the Solid Tumor Evaluation Criteria (RECIST 1.1);
7. Expected survival ≥ 12 weeks;
8. have adequate organ and hematopoietic function, and have laboratory results that meet the requirements

Exclusion Criteria:

in Phase Ia:

* Subjects with any of the following are not eligible for enrollment in this study:

  1. Those who have developed another malignancy within 5 years prior to enrollment, with the exception of cured carcinoma in situ of the cervix and cured basal cell carcinoma of the skin;
  2. Failure to recover from adverse effects of prior therapy to a CTCAE 5.0 grade score of ≤ grade 1, except for residual alopecia areata effects;
  3. Subjects with active, or history of, autoimmune disease with potential for relapse (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or at high risk (e.g., have received an organ transplant requiring immunosuppressive therapy). However, subjects with the following diseases are allowed to enroll:
* Type 1 diabetes mellitus that has stabilized with the use of fixed-dose insulin;
* Autoimmune hypothyroidism requiring only hormone replacement therapy;
* Skin disorders that do not require systemic therapy (e.g., eczema, rashes covering less than 10% of the body surface, psoriasis without ophthalmologic symptoms, etc.); 4) Anticipated major surgery during this study including the 28-day screening period; 5) Subjects requiring treatment with systemic corticosteroids (dose equivalent to >10 mg prednisone/day) or other immunosuppressive medications within 14 days prior to the first dose or during the study period; enrollment is permitted in the following cases:
* Subjects are permitted to use topical topical or inhaled glucocorticoids;
* Short-term (≤ 7 days) use of glucocorticoids for prophylaxis or treatment of non-autoimmune allergic diseases is permitted; 6) Currently suffering from sudden lung disease, interstitial lung disease, interstitial pneumonia, pulmonary fibrosis, acute lung disease, radiation pneumonitis; 7) systemic diseases that have not been controlled and stabilized by treatment, such as cardiovascular diseases (unstable angina pectoris or myocardial infarction before 6 months, etc.) diabetes mellitus, hypertension, etc; 8) arterial or venous thrombosis or embolic events such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months prior to the first dose; 9) History of infection with human immunodeficiency virus, or other acquired, congenital immunodeficiency disease, or history of organ transplantation, or stem cell transplantation; 10) a history of tuberculosis, or a history of tuberculosis disease at the time of screening 11) those with active chronic hepatitis B or active hepatitis C Hepatitis B virus carriers, hepatitis B stabilized by drug therapy (DNA titer must not be higher than 500 IU/mL or copy number <1000copies/ml) and patients with cured hepatitis C (negative HCV RNA test) may be enrolled; 12) Those who have had a serious infection within 4 weeks prior to the first dose or who have had an active infection requiring oral or intravenous antibiotic therapy within the previous 2 weeks;

In phase Ib :

Phase Ib Exclusion Criteria

Subjects with any of the following are not eligible for enrollment in this study:

1. Histologic or pathologic diagnosis of choroidal malignant melanoma;
2. Patients with brain metastases, except those who have been treated and are symptomatically stable. Require ongoing corticosteroids as treatment for CNS disorders, allowing stable doses of anticonvulsant therapy.
3. Malignancies other than malignant melanoma that have occurred within 5 years prior to enrollment, with the exception of malignancies with negligible risk of metastasis or death and/or curative treatment (e.g., adequately treated carcinoma in situ of the cervix, basal or squamous cell skin carcinoma, limited prostate cancer, ductal carcinoma in situ, or stage I uterine cancer);
4. Uncontrolled pleural effusion, abdominal effusion, or pericardial effusion requiring repeated drainage. Those with indwelling drainage tubes are allowed to be enrolled;
5. History of blood transfusion within the last 3 months;
6. hemolytic anemia, autoimmune thrombocytopenia, or Evan syndrome within the last 3 months;
7. prior allogeneic bone marrow transplantation or solid organ transplantation;
8. Failure to recover from adverse effects of prior therapy to a CTCAE 5.0 grade score of ≤ grade 1, excluding alopecia areata;
9. Major surgery within 4 weeks prior to the first dose of study drug or expected to undergo major surgery during the study period;
10. Patients who have received prior CD47 or SIRpa-targeted therapy;
11. have received any live or attenuated vaccine within 28 days prior to the first dose of study drug;
12. have received oral or intravenous antibiotics (including antifungals) 2 weeks prior to the first dose of study drug, except for those who require prophylactic anti-infective therapy (to prevent urinary tract infections or exacerbations of chronic obstructive pulmonary disease);
13. Subjects requiring treatment with systemic corticosteroids (dose equivalent to >10 mg prednisone/day) or other immunosuppressive medications within 14 days prior to the first dose of study drug or during the study period; enrollment is permitted under the following conditions:

    * Use of topical topical or inhaled glucocorticoids;
    * Short-term (≤ 7 days) use of glucocorticoids for prophylaxis or treatment of non-autoimmune allergic diseases;
    * Corticosteroids for the replacement therapy of adrenal insufficiency;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
In phase Ia: Incidence of Dose Limiting Toxicities (DLT) of HX009 in patients with advanced solid tumors | At the end of Cycle 2 (each cycle is 14 days)
  Adverse events (AEs) determined by the investigator are recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0).
Incidence of adverse events (AE) of HX009 in patients with advanced solid tumors | Collected adverse events from signing of informed consent through at least 28 days after the end of treatment, or until other cancer treatment regimens have been started (whichever occurs earlier).
  Adverse events (AEs) determined by the investigator are recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0).
In phase IB:Incidence of Dose Limiting Toxicities (DLT) in HX009 in patients with advanced solid tumors | At the end of Cycle 2 (each cycle is 14 days)
  Incidence and severity of adverse events as assessed by the investigator according to RECIST 1.1;

SECONDARY OUTCOMES:
In Phase Ia: Pharmacokinetics (PK): Maximum plasma concentration of drug (Cmax) | At Cycle 1 ,Cycle 6 and Cycles 2 -5 (each cycle is 14 days)
  Highest concentration of drug measured in the PK samples
Pharmacokinetics (PK): Time to reach Cmax (Tmax) | At Cycle 1 ,Cycle 6 and Cycles 2 -5(each cycle is 14 days)
  Time from dosing until collection of the PK samples with the highest drug concentration.
Terminal Half-life （t½）of HX009 | At Cycle 1 ,Cycle 6 and Cycles 2 -5 (each cycle is 14 days)
  Terminal phase elimination half-life
Area Under the Serum Concentration-time Curve (AUC) | At Cycle 1 ,Cycle 6 and Cycles 2 -5 (each cycle is 14 days)
  The area under the serum concentration-time curve .
Number of Participants With Positive Anti-Drug Antibody (ADA) of HX009 | At Cycles 1-6, 9, 13, 17, and then every 8 cycles up to approximately 1 years: within 1 hour before infusion (each cycle is 14 days).
  ADA blood samples were assayed for anti-HX009 antibodies.
Objective response rate (ORR) of HX009 in patients with solid tumors | Approximately 1 years
  The ORR is defined as the percentage of participants in the analysis population who had a confirmed Complete Response or Partial Response.
Duration of response (DoR) of HX009 in patients with solid tumors | Approximately 1 years
  The DoR is defined as the time from the first recorded response (CR or PR) to the first recorded tumor progression or death due to any cause.
Progression-free survival (PFS) of patients with solid tumors treated with HX009 | Approximately 1 years
  The PFS is defined as the time from the start of the first dose to the first documented disease progression or death of any cause.
In Phase Ib: ORR | Approximately 2 years
  objective response rate assessed by the investigator according to RECIST1.1/iRECIST;
In Phase Ib: DCR | Approximately 2 years
  disease control rate assessed by the investigator according to RECIST1.1/iRECIST;
In Phase Ib: PFS | Approximately 2 years
  progress-freee survival assessed by the investigator according to RECIST1.1/iRECIST;
In Phase Ib: Cmax | Approximately 1 years
  Highest concentration of drug measured in the PK samples
In phase Ib：AUC | Approximately 1 years
  Area Under the Serum Concentration-time Curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciense, Beijing, China

IPD SHARING:
Plan to Share IPD: No